CLINICAL TRIAL: NCT03301870
Title: A Single-Site Study To Evaluate The Irritation Potential Of Topically Applied ATx201 In Healthy Human Volunteers on Intact and Abraded Skin
Brief Title: A Study to Evaluate the Irritation Potential of ATx201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ATx201-006
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Irritation Potential of Topic Agent

STUDY DESIGN:
Intervention Model Description: the assignment of the test articles to the test sites will be randomized. Each "arm" is a different patch of skin on the same study participant
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- ATx201 GEL, 2% - intact skin (Experimental): ATx201 GEL, 2% applied intact skin
  Interventions: Drug: ATx201 Gel 2%
- ATx201 GEL, 4% - intact skin (Experimental): ATx201 GEL, 4% applied to intact skin
  Interventions: Drug: ATx201 Gel 4%
- ATx201 GEL, 2% - abraded skin (Experimental): ATx201 GEL, 2% applied to abraded skin
  Interventions: Drug: ATx201 Gel 2%
- ATx201 GEL, 4% - abraded skin (Experimental): ATx201 GEL, 4% applied to abraded skin
  Interventions: Drug: ATx201 Gel 4%
- ATx201 GEL Placebo - intact skin (Placebo Comparator): ATx201 GEL Placebo applied to intact skin
  Interventions: Drug: ATx201 Placebo
- ATx201 GEL Placebo - abraded skin (Placebo Comparator): ATx201 GEL Placebo applied to abraded skin
  Interventions: Drug: ATx201 Placebo
- Negative Irritant Control - intact skin (Active Comparator): Negative (low) Irritant Control applied to intact skin
  Interventions: Drug: Negative Control
- Negative Irritant Control - abraded skin (Active Comparator): Negative (low) Irritant Control applied to abraded skin
  Interventions: Drug: Negative Control
- Positive Irritant Control - intact skin (Active Comparator): Positive (high) Irritant Control applied to intact skin
  Interventions: Drug: Positive Control

INTERVENTIONS:
Drug: ATx201 Gel 2% — 2% active gel
  Arms: ATx201 GEL, 2% - abraded skin; ATx201 GEL, 2% - intact skin
Drug: ATx201 Gel 4% — 4% active gel
  Arms: ATx201 GEL, 4% - abraded skin; ATx201 GEL, 4% - intact skin
Drug: Positive Control — Sodium Lauryl Sulfate 0.05% (w/v), USP in sterile, distilled Water for Injection, USP
  Arms: Positive Irritant Control - intact skin
Drug: Negative Control — Water for Injection, USP
  Arms: Negative Irritant Control - abraded skin; Negative Irritant Control - intact skin
Drug: ATx201 Placebo — matching placebo gel
  Arms: ATx201 GEL Placebo - abraded skin; ATx201 GEL Placebo - intact skin

SUMMARY:
This is a Phase I single-site study to evaluate the irritation potential of topically applied ATx201 GEL, 2% and 4%, along with positive and negative control and placebo control (ATx201 GEL Placebo), in healthy human subjects on intact and abraded skin. Approximately thirty-six (36) healthy adult subjects will receive all the test articles to provide for 30 subjects to complete the study. The test articles will be applied to the upper back of the subjects during the study, and the placement of the test articles will be randomized. Abraded skin will be induced using sequential tape stripping.

ELIGIBILITY:
Inclusion Criteria:

* Judged by the Investigator to have no health conditions that would impact the safety of the subject during participation.
* Body Mass Index (BMI) to be no less than 19.0 and no greater than 36.0 kg/m² (inclusive).
* Demonstrates a Fitzpatrick skin score of I - IV
* Female subjects must agree to use a medically acceptable contraceptive method
* Willing to refrain from excessive consumption of sodium (> 2,400 mg/day or > 1 teaspoon equivalent/day) in food or beverage 48 hours prior to Day 1 through EOS Visit.
* Willing to shower using the same non-medicated soap/cleansers, and abstain from excessive sun exposure (including tanning salons) from the Screening Visit through EOS Visit.

Exclusion Criteria:

* any clinical investigational product within 30 days prior to Day 1 through EOS Visit
* recent or current medical condition that, in the opinion of the Investigator, might significantly affect an immunological response to topical ATx201 or compromise the safety of the subject.
* history of diabetes mellitus, clinically significant asthma (acceptable if no episode within 5 years prior to Day 1), or currently diagnosed with hypertension or circulatory disease.
* use of any medication on a regular basis within 14 days prior to Day 1 through EOS that could change peripheral blood flow, with the exception of any prescribed birth control method or hormone replacement therapy.
* use of any oral, nasal or topical corticosteroids, or oral or topical retinoids (other than Vitamin A at normal dietary amounts) within 14 days prior to the Screening Visit through EOS Visit.
* intending to start, stop, or change the dose of any prescription or over-the-counter (OTC) medication within 48 hours prior to Day 1 through EOS Visit.
* use of any prescription or OTC topical medications on the upper back within 30 days prior to Day 1 through EOS Visit.
* history of sensitivity/allergy to any ingredients found in the ATx201 formulation or has a history of adverse reactions to topical medications.
* significant history of allergy to soaps, lotions, emollients, ointments, creams, cosmetics, adhesives, or latex.
* history of significant skin conditions or disorders such as psoriasis, atopic dermatitis, etc.
* history of significant dermatologic cancers, for example, melanoma or squamous cell carcinoma.
* displays an obvious difference in skin color on the upper back or the presence of a skin anomaly such as a recent sunburn, scratch, scar tissue, tattoo, or coloration that would interfere with placement of test sites, their assessment, and their potential response to the study drug or that could compromise the safety of the subject.
* smoking or use of tobacco or nicotine delivery products within 14 days prior to Day 1 through EOS Visit.
* female who is pregnant, lactating, breastfeeding, or intends to become pregnant over the course of the study.
* history of drug or alcohol addiction or abuse within the past year.
* caffeine intake greater than 500 mg per day (for example, 1 cup of coffee contains approximately 85 mg of caffeine, tea approximately 25 mg, soft drinks up to 115 mg, energy drinks 90 - 422 mg).
* unwilling to abstain from energy drinks, alcohol, and excessive caffeine (> 500 mg/day) for 48 hours prior to Day 1 through EOS Visit.
* reports having donated blood or plasma within 48 hours prior to Day 1 through EOS Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Cumulative Irritation Scores | 21 days
  the sum of the combined Dermal response and Other Effects Score

SECONDARY OUTCOMES:
Time of combined Dermal response and Other Effects Score >=3 | 21 days
  Total number of days with a combined Dermal Response and Other Effects score of 3 or more for each test article
Incidence of Test Article Discontunation | 21 days
  Number of subjects, by test article, where a test article was discontinued due to an unacceptable degree of irritation, or who experienced symptomatic intolerable irritation
Time to test article discontinuation | 21 days
  Number of days until sufficient irritation occurred to preclude repeat application to the same site, or who experienced symptomatic intolerable irritation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Director — Sponsor CMO
Locations (1):
- Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No